CLINICAL TRIAL: NCT00601692
Title: A Phase I Trial of Irinotecan, Radiation Therapy and Escalating Doses of Docetaxel With Cisplatin in Locally Advanced Esophageal Cancer
Brief Title: Irinotecan, Radiation Therapy, and Docetaxel With or Without Cisplatin in Treating Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02-061; P30CA008748 (NIH); MSKCC-02061; SANOFI-AVENTIS-MSKCC-02061
Record Dates: First submitted 2008-01-17; First posted 2008-01-28 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Esophageal Cancer
Keywords: squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Docetaxel; Irinotecan; Radiotherapy

ARMS (2):
- Regimen 1 (Experimental): Patients receive docetaxel IV over 15 minutes and irinotecan hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 8, patients receive docetaxel IV over 15 minutes and irinotecan hydrochloride IV over 30 minutes on days 1 (week 8) and 8 (week 9). Patients also undergo radiotherapy once daily, 5 days a week, in weeks 8-10. Treatment with chemoradiotherapy repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Regimen 2 (Experimental): Patients receive docetaxel IV and irinotecan hydrochloride as in regimen 1 induction chemotherapy. They also receive cisplatin IV over 20-30 minutes on days 1 and 8. Treatment with irinotecan hydrochloride, docetaxel, and cisplatin repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients receive docetaxel IV, irinotecan hydrochloride IV, and undergo radiotherapy as in regimen 1 chemoradiotherapy. Patients also receive cisplatin IV over 20-30 minutes on days 1 (week 8) and 8 (week 9). Treatment with irinotecan hydrochloride, docetaxel, cisplatin, and radiotherapy repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: irinotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Arms: Regimen 2
Drug: docetaxel — Given IV
Drug: irinotecan hydrochloride — Given IV
Radiation: radiation therapy — Given 5 days a week for 3 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Irinotecan and docetaxel may also make tumor cells more sensitive to radiation therapy. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with irinotecan and radiation therapy with or without cisplatin in treating patients with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose limiting toxicity and recommended phase II dose of docetaxel when given at escalating doses with weekly irinotecan hydrochloride and concurrent radiotherapy in patients with locally advanced esophageal cancer.
* To determine the dose limiting toxicity of cisplatin, once the recommended phase II dose of docetaxel is established, when given weekly with docetaxel, irinotecan hydrochloride, and concurrent radiotherapy in patients with locally advanced esophageal cancer.

Secondary

* To evaluate the clinical and pathological complete response rate in patients with locally advanced esophageal cancer treated with induction chemotherapy comprising docetaxel and irinotecan hydrochloride with or without cisplatin followed by concurrent docetaxel and irinotecan hydrochloride with or without cisplatin plus radiotherapy.

OUTLINE: Patients receive one of the following regimens. Regimen 2 is for patients recruited after the recommended phase II dose has been determined in patients recruited (who receive regimen 1).

* Regimen 1:

  * Induction chemotherapy (weeks 1-6): Patients receive docetaxel IV over 15 minutes and irinotecan hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  * Chemoradiotherapy (weeks 8-13): Beginning in week 8, patients receive docetaxel IV over 15 minutes and irinotecan hydrochloride IV over 30 minutes on days 1 (week 8) and 8 (week 9). Patients also undergo radiotherapy once daily, 5 days a week, in weeks 8-10. Treatment with chemoradiotherapy repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
* Regimen 2:

  * Induction chemotherapy (weeks 1-6): Patients receive docetaxel IV and irinotecan hydrochloride as in regimen 1 induction chemotherapy. They also receive cisplatin IV over 20-30 minutes on days 1 and 8. Treatment with irinotecan hydrochloride, docetaxel, and cisplatin repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  * Chemoradiotherapy (weeks 8-13): Patients receive docetaxel IV, irinotecan hydrochloride IV, and undergo radiotherapy as in regimen 1 chemoradiotherapy. Patients also receive cisplatin IV over 20-30 minutes on days 1 (week 8) and 8 (week 9). Treatment with irinotecan hydrochloride, docetaxel, cisplatin, and radiotherapy repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma, poorly differentiated carcinoma, or carcinoma not otherwise specified, of the esophagus or gastroesophageal (GE) junction

  * Disease clinically limited to the esophagus or GE junction (T1, N1, M0, or T2-4, any N, M0)
  * M1a metastatic disease to lymph nodes allowed

    * Includes celiac lymph nodes in a patient with a distal third esophageal primary lesion or a gastroesophageal junction primary or supraclavicular lymph nodes in a patient with a proximal third esophageal lesion
  * Disease must be able to be contained in a radiotherapy field
* Previously untreated patients with primary tumors of the cervical or thoracic esophagus, including the GE junction, are eligible for this study

  * At least 50% of the tumor must involve the distal esophagus for tumors of the GE junction

Exclusion criteria:

* Positive malignant cytology of the pleura, pericardium, or peritoneum
* Metastatic disease to distant organs (e.g. liver) or non-regional lymph nodes
* Biopsy proven tumor invasion of the tracheobronchial tree or tracheo-esophageal fistula

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status (PS) 70-100% OR ECOG PS 0-2
* ANC ≥ 1,500 cells/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Total serum bilirubin ≤ 1.0 mg/dL
* AST ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Men and women of child bearing potential must use effective contraception while on treatment and for a reasonable period thereafter
* Negative pregnancy test

Exclusion criteria:

* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Pre-existing peripheral neuropathy > grade 1
* Severe comorbid conditions including, but not limited to, any of the following:

  * NYHA class III-IV cardiac disease
  * Myocardial infarction within the past 6 months
  * Severe uncontrolled diabetes
  * Hypercalcemia
  * Uncontrolled hypertension
  * Cerebral vascular disease
  * Uncontrolled infections
* Pregnant or lactating women
* History of prior malignancy diagnosed and/or treated within the past three years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or superficial transitional cell carcinoma of the bladder
* Known Gilbert disease
* History of seizure disorder with concurrent phenytoin, phenobarbital, or other antiepileptic medication
* Any other concurrent medical or psychiatric condition or disease that, in the investigator's judgment, would make the patient inappropriate for entry into this study
* Patients who cannot fully comprehend the therapeutic implications of the protocol or comply with the requirements

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy (RT) for this esophageal cancer
* No prior mantle RT, chest RT, pelvic RT, or hemi-body RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of docetaxel when administered together with irinotecan hydrochloride and radiotherapy | 2 years

SECONDARY OUTCOMES:
Clinical and pathological complete response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States